CLINICAL TRIAL: NCT06244225
Title: An Exploratory Study to Evaluate the Efficacy and Safety of Hepatic Arterial Infusion Chemotherapy (HAIC) Combine With Sintilimab and Donafenib for Unresectable Hepatocellular Carcinoma
Brief Title: HAIC (Hepatic Artery Infusion Chemotherapy，HAIC）Plus Sintilimab and Donafenib in the First-line Treatment of Unresectable Hepatocellular Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UHCT230851
Record Dates: First submitted 2024-01-29; First posted 2024-02-06 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-01

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HAIC + Sintilimab + Donafenib (Experimental): HAIC combine with Sintilimab and Donafenib
  Interventions: Drug: Donafenib； Sintilimab； HAIC

INTERVENTIONS:
Drug: Donafenib； Sintilimab； HAIC — Drug: Sintilimab Q3W 200mg IV d1, Q3W
  Drug: Donafenib 200 mg BID d1-21, Q3W
  other: HAIC Q3W Oxaliplatin: 85mg/m2 , Day 1 Leucovorin: 200mg/m2, Day 1 Fluorouracil: 400mg/m2, Day1 and 2400mg/m2 continuous arterial perfusion for 46h.

SUMMARY:
This is a single-arm exploratory clinical study to evaluate the efficacy and safety of HAIC in combination with Sintilimab and Donafenib in patients with BCLC-C stage who have not received prior systemic therapy

DETAILED DESCRIPTION:
This trial is a single-arm, non-randomized and single-center clinical study of HAIC in combination with Sintilimab and Donafenib in the first-line treatment of BCLC-C stage unresectable hepatocellular carcinoma. The study is expected to include 38 subjects who meet the screening criteria to receive HAIC plus Sintilimab and Donafenib to evaluate the efficacy and safety of treatment, including time to progression（PFS）and overall survival（OS），etc.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent should be signed before implementing any trial-related procedures
2. ECOG PS scores 0-1
3. Histologically/cytologically confirmed HCC or cirrhosis meeting the clinical diagnostic criteria of HCC by American Association for the Study of Liver Diseases (AASLD)
4. Barcelona Clinic Liver Cancer (BCLC) stage C
5. Newly diagnosed HHC patients without any previous treatment for the tumor
6. Child Pugh score of ≤ 7.
7. Estimated survival > 12 weeks
8. At least one measurable lesion according to RECIST V1.1
9. Sufficient organ and bone marrow functions

Exclusion Criteria:

1. Histologically/cytologically confirmed fibrolamellar hepatocellular carcinoma, sarcomatoid hepatocellular carcinoma, and cholangiocarcinoma.
2. History of hepatic encephalopathy or liver transplantation.
3. Symptomatic pleural effusion, ascites, and pericardial effusion that require drainage.
4. Acute or chronic active hepatitis B or C infection; hepatitis B virus (HBV) DNA > 2000 IU/mL or 104 copies/mL; hepatitis C virus (HCV) RNA > 103 copies/mL; hepatitis B surface antigen (HbsAg) and anti HCV antibody positive concurrently.
5. Presence of metastasis to the central nervous system.
6. Presence of bleeding events from esophageal or gastric varices caused by portal hypertension within the past 6 months. Presence of known severe (G3) varicose veins in endoscopy within 3 months before the first dose. Evidence of portal hypertension (including the finding of splenomegaly in imaging studies) with a high risk of bleeding assessed by the investigator.
7. Presence of any life-threatening bleeding events within the past 3 months, including the need for transfusion, surgery or local treatment, and continuous medication therapy.
8. Any arterial/venous thromboembolic events within 6 months, including myocardial infarction, unstable angina, cerebrovascular accident or transient cerebral ischemic attack, pulmonary embolism, deep vein thrombosis, or any other history of serious thromboembolism. Presence of implantable venous port or catheter derived thrombosis, or superficial venous thrombosis, barring stable thrombosis following the conventional anticoagulation treatment. Prophylactic use of low dose low molecular weight heparin (e.g., enoxaparin 40 mg/day) is permitted.
9. Involvement of both the main portal vein and the left and right branches by portal vein tumor thrombus, or of both the main trunk and the superior mesenteric vein concurrently. Presence of tumor thrombus of inferior vena cava.
10. A 10-day consecutive dosing of aspirin (> 325 mg/day) or other drugs, e.g., dipyridamole and clopidogrel, known to inhibit the platelet function within 2 weeks before the first dose.
11. Uncontrolled hypertension (systolic greater than 140 mmHg or diastolic greater than 90 mmHg) after the optimal medical treatment, history of hypertensive crisis or hypertensive encephalopathy.
12. Toxicity (excluding alopecia, events not clinically significant, and asymptomatic laboratory abnormalities) caused by previous therapy that has not yet resolved to grade 0 or 1 (National Cancer Institute Common Terminology Criteria for Adverse Events V5.0 (NCI CTCAE V5.0)) before the first dose of study drugs.
13. Symptomatic congestive cardiac failure (NYHA Class II IV). Symptomatic or poorly controlled arrhythmia. History of congenital long QT syndrome or corrected QTc > 500 ms (calculated using Fridericia formula) during screening.
14. Serious hemorrhagic tendency or coagulopathy, or currently receiving thrombolytic therapy.
15. History of gastrointestinal perforation and/or fistula, history of bowel obstruction (including incomplete bowel obstruction requiring parenteral nutrition), extensive bowel resection (partial colectomy or extensive small bowel resection accompanied with chronic diarrhea), Crohn's disease, ulcerative colitis, or chronic diarrhea within the past 6 months.
16. Receipt of immunosuppressants within 4 weeks before the first dose, excluding local glucocorticoids administered by nasal, inhaled, or other topical routes, or systemic glucocorticoids of physiological doses (no more than 10 mg/day of prednisone or equivalents), while the temporary use of glucocorticoids for preventing allergies or treating dyspneic symptoms of such diseases as asthma and chronic obstructive pulmonary disease is permitted.
17. Receipt of a live attenuated vaccine within 4 weeks before the first dose or planned to receive a live attenuated vaccine during the study.
18. Receipt of major surgery (craniotomy, thoracotomy, or laparotomy) within 4 weeks before the first dose or having unhealed wounds, ulcers, or fractures. Receipt of tissue biopsy or other minor surgeries within 7 days before the first dose, barring venipuncture and catheterization for intravenous infusion.
19. Receipt of local treatment for liver cancer within 4 weeks before the first dose.

    Receipt of systemic treatment with traditional Chinese medicines with cancer indications or immunomodulators (including thymosin, interferon, and interleukin, barring local use for controlling pleural fluid or ascites) within 2 weeks before the first dose.
20. Uncontrolled/uncorrectable metabolic disorders, other non malignant organ diseases, systemic diseases, or cancer related secondary diseases with the potential to cause a relatively high medical risk and/or survival evaluation uncertainties unsuitable for subject enrollment as judged by the investigator; other circumstances unsuitable for subject enrollment as judged by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) per RECIST v1.1 | From baseline to primary completion date, about 18 months
  Defined as a duration from the date of initial treatment to disease progression or death of any cause

SECONDARY OUTCOMES:
Overall response rate (ORR) per RECIST v1.1 and mRECIST | From baseline to primary completion date, about 18 months
  Defined as the incidence of complete response and, partial response
Disease control rate (DCR) per RECIST v1.1 and mRECIST | From baseline to primary completion date, about 18 months
  Defined as the incidence of complete response, partial response and stable disease
Overall survival (OS) | From baseline to primary completion date, about 18 months
  Defined as a duration from the date of initial treatment to death of any cause.
Duration of response (DoR) per RECIST v1.1 and mRECIST | From baseline to primary completion date, about 18 months
  Defined as a duration from date of initial treatment to disease progression or death in patients who achieve complete or partial response
The treatment-related adverse events (TRAEs） | From baseline to primary completion date, about 18 months
  Defined as the proportion of patients with AE, treatment-related AE (TRAE), immune-related AE (irAE), serious adverse event (SAE), assessed by NCI CTCAE v5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Union Hospital affiliated to Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No